CLINICAL TRIAL: NCT01575951
Title: Pilot Study: Dynamic Contrast-enhanced Magnetic Resonance Imaging(DCE-MRI)for Assessing Tumor Vascularity and Permeability in Soft Tissue Sarcoma Treated With Preoperative Radiotherapy Followed by Surgical Resection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HCI38583
Record Dates: First submitted 2012-01-30; First posted 2012-04-12 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental): All participants enrolled.
  Interventions: Radiation: MRI-DCE

INTERVENTIONS:
Radiation: MRI-DCE — The treatment follows the standard practice including radiation dose and treatment volumes.
  DCE-MRI imaging is to be performed immediately after CT simulation using the same immobilization device.
  Pre-op DCE-MRI is performed and integrated into radiation simulation planning which is considered a standard technique for radiation oncologist to assess tumor volume and peritumoral edma. It will make radiation field more accurate and precise. This MRI is to be performed on the date of simulation immediately after CT simulation.
  MRI image data is then transferred into radiation eclipse system, and integrated into the planning system for target contouring.
  Follow the standard pre-operative radiotherapy technique using 3D conformal radiotherapy (3DCRT) or intensity modulated radiation therapy (IMRT) to deliver a total dose of 50 Gy at 2 Gy per fraction for trunk or extremity STS, or 45 Gy at 1.8 Gy per fraction for retroperitoneal STS, 5 treatments per week.

SUMMARY:
This is a pilot study to determine the diagnostic value of dynamic contrast enhancing MRI (DCE-MRI) in soft tissue sarcoma for assessment of tumor radiographic changes in vascular permeability and microvessel density before and after preoperative radiotherapy.

DETAILED DESCRIPTION:
All patients have biopsy proven soft tissue sarcoma and undergo preoperative radiotherapy. Dynamic contrast-enhancing MRI T1-weight DCE-MRI will cover the whole tumor and involved lymph nodes if indicated. DCE-MRI is obtained before radiation starts and 4 weeks after RT completes. Blood volume images are estimated by using general Toft model, by which the blood flow was corrected for vascular permeability and perfusion. These images are geometrically co-registered with post-Gd T1-weighted MR images and pre-op RT routine MRI images are fused with the treatment planning CT.

Routine and DCE-MRI will be evaluated in each patient to determine the gross tumor volume. The quantitative parameters are determined on DCE-MRI for quantitative parameters in blood flow and permeability in the region of interest. Dynamic images are converted into color maps reflecting Ktrans, kep, Ve, and mean value of each parameter.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed soft tissue sarcoma.
2. Age ≥ 18.
3. ECOG 0-1.
4. Able to receive preoperative radiotherapy followed by surgical resection.
5. Able to provide treatment consent forms that conforms to federal and institutional guidelines.
6. Have adequate kidney function for safe administration of gadolinium contrast, as determined by current Department of Radiology MRI guidelines.
7. Creatinine clearance either by 24 hour collection or nomogram:

Creatinine clearance (CC) > 50 ml/min is determined by 24 hour collection or nomogram: CC male = (140 - age) x (wt. in kg)/(Serum Cr mg/dl) x 72 CC female = 0.85 x (CC male)

Exclusion Criteria:

1. Patients have claustrophobia, iron or metal in the MRI scan site or pacemaker which are contraindicated for MRI scan.
2. patients have pacemaker or defibrillator and contraindicated to MRI images
3. Patients are allergic to gadolinium IV contrast.
4. Patients have acute or chronic renal insufficiency and contraindicated to gadolinium contrast enhancing MRI.
5. Patient had previous radiation to the same disease site.
6. Patient had chemotherapy prior to preoperative radiotherapy.
7. Patients that are pregnant. Patients that may become pregnant must have a negative pregnancy test prior to enrolling.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-02; Primary Completion 2014-11-05 (Actual); Study Completion 2014-12-05 (Actual)

PRIMARY OUTCOMES:
Feasibility | 36 months
  Feasibility of DCE-MRI (Dynamic contrast-enhancing) in adult soft tissue sarcoma

SECONDARY OUTCOMES:
Necrosis level | 36 months
  We will measure necrosis within the ROI (region of interest).
Tumor Volume change | 36 months
  We will measure tumor volume change of tissues within the ROI (region of interest).

CONTACTS AND LOCATIONS:
Overall Officials: Ying Hitchcock, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States